CLINICAL TRIAL: NCT06245252
Title: Comparison of Passive Stretching Versus Electrical Stimulation on Glucose Level, Functional Mobility and Perceived-fatigue in Elderly With Type II Diabetes
Brief Title: Passive Stretching Versus Electrical Stimulation on Glucose Level, in Elderly With Type II Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mona Mohamed Abdelkhalek (Other)
Responsible Party: Sponsor-Investigator, Mona Mohamed Abdelkhalek, assistance professor, Badr University
Organization: Badr University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mona 1
Record Dates: First submitted 2023-12-19; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Type II Diabetes
Keywords: blood glucose; electrical stimulation; lower extremities; passive stretching; exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Muscle Stretching Exercises; Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (A) (Experimental): treated by 40-minute passive stretching exercises,three times per week for 12 weeks
  Interventions: Other: passive stretching for group A
- group (B) (Experimental): treated by 30 minutes electrical stimulation three times per week for 12 weeks
  Interventions: Other: electrical stimulation for group b

INTERVENTIONS:
Other: passive stretching for group A — A description of stretch is performed 3 times per week for 12 weeks. The stretches included (in the order they were applied): Seated knee flexor (bilateral); Seated knee flexor-hip adductor (bilateral); Seated shoulder lateral flexor (bilateral); Supine hip flexor- knee extensor (unilateral). Seated hip external rotators, extensor (unilateral); Seated shoulder extensors, adductors, retractors (unilateral). Supine knee flexor-plantar flexor (unilateral); Prone hip flexor (unilateral); Seated shoulder flexors, depressors (bilateral); Seated shoulder and elbow flexors (unilateral).
  Other Names: passive stretching exercises for group A
  Arms: group (A)
Other: electrical stimulation for group b — reated by 30 minutes electrical stimulation three times per week for 12 weeks
  Arms: group (B)

SUMMARY:
Sixty elderly diabetics (type II) their age ranged from 60-75 years had been divided into two equal groups; group (A) treated by 40-minute passive stretching exercises, while the group (B) treated by 30 minutes electrical stimulation three times per week for 12 weeks. Blood glucose level,Time up and go test (TUG) and Fatigue severity scale were done before and after 12 weeks of the study.Conclusion: Both electrical stimulation and passive stretching are effective to lowering blood glucose level and can be proposed for those people restricted to perform exercise.

DETAILED DESCRIPTION:
Background: Physical exercise is one of the bases for controlling and treatment type 2 diabetes mellitus. But not all diabetic elderly is able to perform physical exercise because of their physical limitation condition. The approach for those people in this study is electrical stimulation and passive stretching. Purpose: The aim of this study is to compare the effect of passive stretching and electrical stimulation on blood glucose level, functional mobility and Perceived-Fatigue in diabetic elderly. Methods: Sixty elderly diabetics (type II) their age ranged from 60-75 years had been divided into two equal groups; group (A) treated by 40-minute passive stretching exercises, while the group (B) treated by 30 minutes electrical stimulation three times per week for 12 weeks. Blood glucose level,Time up and go test (TUG) and Fatigue severity scale were done before and after 12 weeks of the study.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c value between 6.5% -8.5%,
* age ranged from 60-75 years patients have
* body mass index (BMI) from 25 to 29.9 kg/m2,
* duration of diabetes ranged from 5-7 years. They were
* on oral hypoglycemic medications at the same dose.
* All patients were clinically and medically stable when attending the study.

Exclusion Criteria:

* unstable cardiovascular,
* chest problems
* other types of diabetes
* on insulin therapy
* chronic renal failure and
* iron deficient anemia and
* musculoskeletal disorders which may affect their physical ability to do the exercises.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-10 (Estimated); Primary Completion 2024-05-10 (Estimated); Study Completion 2024-06-10 (Estimated)

PRIMARY OUTCOMES:
an HbA1c . | at baseline and after three month
  blood glucose levels glycated haemoglobien
fasting blood glucose levels | at baseline and after three month
  values were obtained for fasting blood sugar (FBS) levels/baseline, then 2 hours after the meal (postprandial).

SECONDARY OUTCOMES:
time of up and go test | at baseline and after three month
  measure the time of the test
score of fatigue severity scale | at baseline and after three month
  severity from 1 to 7The strongly disagreement was related to number 1 while the strongly agreement was related to number 7. The scoring is completed by calculating the average answer to the questions (adding up all the answers and dividing by nine). Greater FSS scores mean greater perceived-fatigue.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Badr university, Cairo
  - Mona Mohamed Abdelkhalek, Cairo